CLINICAL TRIAL: NCT07186283
Title: A Phase 1 Study to Assess the Safety and Pharmacokinetics of Novel Cannabidiol (CBD) Soft-gel Capsule Formulation (NW300EMCBD) in Healthy Subjects
Brief Title: Pharmacokinetic Study of a Novel Cannabidiol (CBD) Formulation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NW PharmaTech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NWPharma_CH_001
Record Dates: First submitted 2025-09-05; First posted 2025-09-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: PK in Healthy Volunteers
Keywords: Cannabidiol formulation; Cannabidiol pharmacokinetic; Encapsulated Micellar CBD formulation; Cannabidiol safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NW300EMCBD 600 mg (Experimental): 600 mg CBD soft-gel capsules (novel formulation)
  Interventions: Drug: CBD soft-gel capsules 600 mg
- NW300EMCBD 900 mg (Experimental): 900 mg CBD soft-gel capsules (novel formulation)
  Interventions: Drug: CBD soft-gel capsules 900 mg
- Epidyolex (Active Comparator): 25 mg/kg
  Interventions: Drug: Epidyolex

INTERVENTIONS:
Drug: CBD soft-gel capsules 600 mg — 600 mg
  Arms: NW300EMCBD 600 mg
Drug: CBD soft-gel capsules 900 mg — 900 mg
  Arms: NW300EMCBD 900 mg
Drug: Epidyolex — 25 mg/kg
  Arms: Epidyolex

SUMMARY:
The purpose of this study is to test a new formulation of cannabidiol (CBD) to see how it is processed in the body and how safe it is for healthy volunteers. CBD is a compound found in the cannabis plant that has shown potential to help treat various medical and mental health conditions. While there is already an approved CBD-based drug that is used for epilepsy in the UK, called Epidyolex, most CBD formulations have poor absorption when taken orally, reducing their effectiveness and often requiring higher doses.

NW PharmaTech has developed a new CBD formulation aimed at improving absorption and processing by the body. This study will assess the absorption, safety, and tolerability of two different doses (600 mg and 900 mg) of the new formulation and will compare them with Epidyolex (dosed as per approved label).

All participants will receive each of the following three dosing regimens in a randomised order across three separate experimental periods, with each period separated by a 25 day washout period, which ensures that the drug from one dosing regimen is fully cleared from your body before the next dosing regimen begins.

Regimen A: 600 mg of the new CBD formulation (NW300EMCBD) administered orally Regimen B: 900 mg of the new CBD formulation (NW300EMCBD) administered orally Regimen C: 25 mg/kg Epidyolex solution (2 x 12.5 mg/kg doses separated by 12 hours) administered orally In total, participants will complete three dosing visits (one per experimental period), each spaced 25 days apart. The study will evaluate the pharmacokinetics (PK) of the formulations, which refers to how the body absorbs, distributes, metabolizes, and eliminates the drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers.
2. Age range between 18 and 55 years old.
3. Weight at least 50kg and have a body mass index (BMI) between 19 and 30 kg/m2 at screening.
4. Willingness to comply with and complete all study procedures, including consuming the protocol specified high-fat, high-calorie meal in 30 minutes.
5. In good health, as determined by no clinically significant findings from medical history, 12-lead ECG and vital signs measurements, and clinical laboratory evaluations at screening and check-in, and from the physical examination at screening and symptom-directed physical examination at baseline, as assessed by the investigator or designee.
6. Abstinence from consuming St John's wort, grapefruit (juice), alcohol or tobacco and nicotine products for at least 72 hours prior to dosing and throughout treatment period.
7. Abstinence from caffeine for the duration of the in-clinic confinement period, including all dosing days. Caffeinated beverages and products will not be available on site.
8. Capable and willing to comply with protocol requirements during the study.
9. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Participation in a research clinical trial within 90 days prior to Day 1 of the first experimental period, or 5 elimination half-lives prior to Day 1 of the first experimental period (whichever is longer) to Day 1, or throughout the study.
2. Use of cannabis products, including hemp, in any form (including medication, oils, edibles or drinks) during the last 28 days before screening.
3. History of hypersensitivity or allergy to CBD oil, sesame oil, hemp or any other cannabinoid products, or any of the items that could be included in the standardized meals/snacks.
4. Using any regular medication in the 28 days prior to screening and throughout the study (as required doses of paracetamol or non-steroidal anti-inflammatory drugs (NSAIDs) are permitted).
5. Abnormal screening sample: clinically significant liver, renal or haematological abnormalities, including total Bilirubin, ALT or AST > the upper limit of normal (ULN).
6. Positive screening test indicating active infection with HIV, hepatitis B virus or hepatitis C virus. Participants with evidence of past HBV infection and complete recovery may be eligible, at the discretion of the Investigator, provided liver function tests are within normal limits and there is no evidence of active infection.
7. Positive urine drug sample, including THC, at screening and, baseline excluding THC at post-dose.
8. Positive alcohol breathalyser test at screening and throughout the study.
9. Any suicidal ideation or behaviour in the past 12 months as assessed by responses to Columbia Suicidal Severity Rating questionnaire at screening.
10. Any history of mental disorder including major depressive disorder, bipolar disorder, psychosis, and any current substance use disorder, including alcohol and tobacco use disorder.
11. Any self-reported, observed or assessed medical condition that might put the subject at risk according to the physician's opinion.
12. Any significant previous or current history of comorbidities capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data.
13. Participants with a sitting blood pressure at screening, after resting for 5 minutes, higher than 140/90 mmHg or lower than 90/50 mmHg.
14. Blood donation or loss (eg surgery) over 200 ml in 3 months prior to screening and throughout study (menstruation is acceptable).
15. Male participants not willing to use contraceptive methods throughout the study.
16. Female participants who are pregnant (positive B-hCG urine test), lactating or breastfeeding.
17. Female participants of childbearing potential* and not willing to use highly effective contraceptive methods** at screening or throughout the study.

    *Defined as females who have experienced menarche and are not surgically sterilised (eg hysterectomy, bilateral salpingectomy) or post-menopausal.

    **Highly effective methods of birth control are those with a failure rate <1% per year and include combined oestrogen and progesterone hormonal contraception, progestogen-only hormonal contraception, intrauterine devices (IUD), intrauterine hormone-releasing systems (IUS) and vasectomised partner.
18. Participants with planned surgical or medical treatment requiring hospitalisation during the study.
19. Employees or family members of the Sponsor.
20. Participant unable to communicate reliably with research team.
21. Participant is not able to swallow capsules.
22. Subject unable or unwilling to consume the protocol specified high fat meal required by the trial protocol and/or the soft gel capsules, which contain gelatine of bovine origin, and/or Epidyolex which contains sesame oil and ethanol.
23. Subjects with alcohol consumption > 14U/ week.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
CBD plasma concentration | Pre-dose up to 192 hours post dose
  Difference in CBD plasma concentration between the novel formulation and Epidyolex

SECONDARY OUTCOMES:
Total Area Under the Curve (AUCinf) | Pre-dose up to 192 hours post dose
  Difference in CBD total exposure between the novel formulation and Epidyolex
Total Area Under the Curve (AUCt) | Pre-dose up to 192 hours post dose
  Difference in CBD total exposure between the novel formulation and Epidyolex
Dose-normalised Total Area Under the Curve (AUCinf/D) | Pre-dose up to 192 hours post dose
  Difference in CBD total exposure normalised by administered CBD total dose between the novel formulation and Epidyolex
Cmax | Pre-dose up to 192 hours post dose
  Maximum plasma concentration
Tmax | Pre-dose up to 192 hours post dose
  Time to reach maximum plasma concentration
Plasma Half-life (t½) | Pre-dose up to 192 hours post dose
  Time to reduce the plasma concentration by half
Apparent plasma clearance (CL/F) | Pre-dose up to 192 hours post dose
Apparent volume of distribution (Vz/F) | Pre-dose up to 192 hours post dose
Elimination rate constant (Kel) | Pre-dose up to 192 hours post dose
Number of participants with Adverse Events (AEs) | Pre-dose up to 192 hours post dose
Changes from pre-dose baseline in laboratory findings | Pre-dose up to 192 hours post dose
  laboratory sampling
Changes from pre-dose baseline Blood Pressure (BP) | Pre-dose up to 192 hours post dose
Changes from pre-dose baseline in Heart Rate (HR) | Pre-dose up to 192 hours post dose
Changes from pre-dose baseline in vital signs Respiratory Rate | Pre-dose up to 192 hours post dose
Changes from pre-dose baseline in Body Temperature | Pre-dose up to 192 hours post dose
Number of participants with ECG findings | Pre-dose up to 192 hours post dose
Changes from pre-dose baseline iGastrointestinal Symptom Rating Scale (GSRS) score | Pre-dose to 24 hours post dose
  The GSRS is a 15-item rating scale, where each item is assessed with a 7-point Likert scale, with higher scores indicating more severe symptoms.
Number of participants with suicidal ideation and/or behavior as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Pre-dose up to 192 hours post dose
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician administered assessment tool that evaluates suicidal ideation and behavior. Number of participants that have an affirmative response provided to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 6 items for suicidal behavior (1. Actual attempt, 2. Interrupted attempt, 3. Aborted attempt, 4. Preparatory acts or behavior, 5. Suicidal Behavior 6. Completed suicide,) will be reported.

OTHER OUTCOMES:
Change in VAMS subscales (mental sedation subscale, tranquilisation and calming effects subscale, physical sedation subscale, other feelings and effects subscale) | Pre-dose to 3 hours post dose
  The Visual Analog Mood Scale (VAMS) measures subjective mood states. Participants mark their feelings on a 100-mm line, scored from 0 (not at all) to 100 (extremely). For the subscales (Mental Sedation, Tranquilization and Calming Effects, Physical Sedation, Other Feelings and Effects), higher scores indicate greater intensity of the measured effect.
Change in the Drug Experience Questionnaire (DEQ-5) | Pre-dose to 3 hours post dose
  The DEQ-5 is a brief self-report measure designed to assess acute subjective experiences of drug effects. It comprises five items in which participants rate their current experiences of drug effect, feeling "high," liking the drug effects, disliking the drug effects, and wanting more of the substance. Responses are recorded using 100-mm visual analog scales, scored from 0 (not at all) to 100 (extremely). Higher scores indicate greater intensity of the subjective experience being measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea Clinical Research Unit (Drapers Yard), Leeds, West Yorkshire, United Kingdom